CLINICAL TRIAL: NCT02859532
Title: Study of Elastographic Properties of the Clot by Technical SWIRE (Shear Wave Induced Resonance Elastography)
Acronym: ClotStruct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.355
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Deep Vein Thrombosis
Keywords: blood coagulation; Endogenous Thrombin Potential; rotational thromboelastometry
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis of deep vein thrombosis (Experimental): All subjects with proximal DVT will have quantitative elastography SWIRE, thrombin generation test and rotational thromboelastometry test.
  Interventions: Radiation: elastography SWIRE

INTERVENTIONS:
Radiation: elastography SWIRE
  Other Names: Supersonic Imagine

SUMMARY:
Deep vein thrombosis (DVT) is a vascular disease characterized by the formation of a thrombus within the venous system, mainly the lower limbs. The clot structure directly influences both its location, but also its progressive profile expansion material or regression and embolic migration.

Few data are available regarding the evolution of structural properties of thrombus after an acute episode of DVT. Thrombus formation is due to the polymerization of fibrinogen into fibrin. Fibrin is a viscoelastic polymer. Its mechanical properties directly determine how the thrombus responds to forces which it is subjected.

Determining the mechanical properties of the thrombus in vivo and ex vivo is expected to study its evolutionary properties.

DETAILED DESCRIPTION:
The main objective of the study is to characterize the in vivo properties of elastographic thrombus in patients with proximal deep vein thrombosis (DVT), for quantitative elastography performed at D0, D7, D30.

The ability to analyze the structural properties of the thrombus should allow us to then correlate these properties to the evolving nature of the thrombus (embolic migration or not, recanalization or not), and the effect of different treatment on the evolution of the thrombus

ELIGIBILITY:
Inclusion Criteria:

* Patient with proximal DVT, provoked or not, the symptomatology is less than 3d, with or without pulmonary embolism treated with heparin or oral anticoagulant
* Signed informed consent
* Patient affiliated to a social security scheme,

Exclusion Criteria:

* pregnant or lactating
* Life expectancy <1 month
* Patient with distal DVT or asymptomatic DVT accidental discovery
* Patient who underwent venous unclogging in acute phase
* exclusion period in another study,
* under administrative or judicial oversight, under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in in vivo elastographic properties of thrombus in patients with proximal deep vein thrombosis (DVT) through quantitative elastography | Day 0, Day 7, Day 30

SECONDARY OUTCOMES:
Thrombus properties depending on the existence or absence of pulmonary embolism (PE) associated | Day 0, Day 7, Day 30
Thrombus properties if provoked versus unprovoked thrombosis | Day 0, Day 7, Day 30
Correlation of the thrombus in vivo properties to the thrombin generation capacity and viscoelastic properties tested ex vivo by rotational thromboelastometry | Day 0, Day 7, Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Gilles PERNOD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No